CLINICAL TRIAL: NCT04282148
Title: A Clinical Investigation to Assess the Abbott Next Generation Drug Eluting Stent 48mm Everolimus Eluting Coronary Stent System (EECSS) in Treatment of de Novo Native Coronary Artery Disease
Brief Title: Abbott Next Generation Drug Eluting Stent 48mm Study
Acronym: SPIRIT 48
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10321
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
Keywords: De novo native coronary artery long lesions; ABT NG DES 48 EECSS; ABT-CIP-10321; Coronary artery luminal diameter; SPIRIT 48
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, global (US and OUS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ABT NG DES 48 EECSS (Experimental): Participants will receive ABT NG DES 48 EECSS device
  Interventions: Device: ABT NG DES 48 EECSS

INTERVENTIONS:
Device: ABT NG DES 48 EECSS — Each participant will receive ABT NG DES 48 EECSS with appropriate diameter

SUMMARY:
The purpose of this SPIRIT 48 study is to evaluate the safety and effectiveness of the ABT NG DES 48 in improving coronary artery luminal diameter in subjects with coronary artery disease (CAD) due to de novo native coronary artery long lesions.

DETAILED DESCRIPTION:
The SPIRIT 48 mm study is a prospective, single arm, open-label, multi-center global (US and outside of US) clinical investigation to evaluate the safety and effectiveness of the ABT Next Generation Drug Eluting Stent 48 mm everolimus-eluting coronary stent system (EECSS) (called "ABT NG DES 48") in up to 107 subjects at up to 33 sites globally. The clinical outcomes from the SPIRIT 48 study will be compared to a performance goal (PG) established using historical control data from the SPIRIT Prime Long Lesion Registry. This clinical investigation will be conducted under an investigational device exemption (IDE) and is intended to support market approval of the ABT NG DES 48 in the United States.

ELIGIBILITY:
General Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedure, per site requirements.
3. Subject must have evidence of myocardial ischemia (e.g., unstable angina, post-infarct angina, stable angina or silent ischemia) suitable for non-emergent PCI. Subject with stable angina or silent ischemia must have objective sign of ischemia as suggested by one of the following,

   * Abnormal stress or imaging stress test
   * Abnormal computed tomography-fractional flow reserve (CT-FFR)
   * Stenosis by visual estimation ≥ 70%
   * Abnormal pressure-derived indexes (FFR, instantaneous wave-free ratio [iFR], or relative flow reserve [RFR])
4. Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Subject must agree not to participate in any other clinical study for a period of one year following the index procedure.

Angiographic Inclusion Criteria:

1. Only one de novo target lesion in native coronary artery is allowed to be treated with the investigational stent.

   • One additional non-target lesion can be treated if it is located in a different epicardial coronary vessel and NOT in left main coronary artery. The non-target lesion must be treated first and must be deemed an angiographic success.
2. The target lesion must be located in a native coronary artery with:

   * Visually estimated reference vessel diameter (RVD) of ≥ 2.5 mm and ≤ 4.25 mm.
   * Visually estimated lesion length of > 32 mm and ≤ 44 mm, and able to be covered by a single ABT NG DES 48.

     a. Multiple focal de novo lesions in an epicardial coronary vessel are allowed if the lesions can be covered by one stent. Multiple focal de novo lesions will be counted as a single lesion.
   * Visually estimated diameter stenosis of > 50% and < 100% with a Thrombolysis in Myocardial Infarction (TIMI) flow of ≥ 1

     1. Stable angina or silent ischemia subjects must have stenosis ≥ 70%, or abnormal pressure-derived physiological indices (FFR, iFR, or RFR), unless abnormal stress or imaging stress test is evidenced.

General Exclusion Criteria:

1. Subject has known hypersensitivity or contraindication to device material and its degradants (everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoropolymers, etc.), or has known contrast sensitivity.
2. Subject has known hypersensitivity or contraindication to aspirin, heparin/bivalirudin, P2Y12 inhibitors (clopidogrel /prasugrel /ticagrelor), and therefore cannot be adequately pre-medicated.
3. Subject has a planned surgery or procedure necessitating discontinuation of aspirin or P2Y12 inhibitor within 12 months following index procedure.
4. Subject is receiving or will require chronic anticoagulation therapy (e.g., coumadin, dabigatran, apixaban, rivaroxaban or any other agent for any reason).
5. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.
6. Subject had an acute myocardial infarction (AMI) within 48 hours of the index procedure with either of the situations below:

   * The subject is currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate-unresponsive prolonged chest pain with ischemic electrocardiogram (ECG) changes
   * Elevated cardiac biomarker values have not returned to within normal limits at the time of index procedure.
7. Subject has a left ventricular ejection fraction (LVEF) < 30% within 3 months prior to the index procedure, that was documented by any method.
8. Subject is expected to require percutaneous mechanical cardiac support at the index procedure.
9. Prior PCI within the target vessel during the last 12 months prior to consent.
10. Prior PCI within the non-target vessel or any peripheral intervention during the last 30 days prior to consent.
11. At the index procedure, subject is identified to require planned stenting procedure (including staged procedures) or CABG after the index procedure.
12. Subject has received a solid organ transplant which is functioning or is active on a waiting list for any solid organ transplants with expected transplantation within 24 months.
13. Subject has a malignancy that is not in remission.
14. Subject is receiving immunosuppressant therapy or has known life-threatening immunosuppressive or severe autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.). Note: corticosteroids are not included as immunosuppressant therapy, diabetes mellitus is not regarded as autoimmune disease
15. Subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy), or the chest/mediastinum.
16. Subject has a platelet count < 100,000 cells/mm^3 or > 700,000 cells/mm^3.
17. Subject has renal insufficiency as defined as an estimated glomerular filtration rate (GFR) < 30 ml/min/1.73m^2 or dialysis at the time of consent.
18. Subject is high risk of bleeding for any reason; has a history of bleeding diathesis or coagulopathy; has had a significant gastro-intestinal or significant urinary bleed within the past six months.
19. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past 6 months, or any prior intracranial bleed, or any permanent neurologic defect, or any known intracranial pathology (e.g. aneurysm, arteriovenous malformation, etc.).
20. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion. Note: femoral arterial disease does not exclude the subject if radial access may be used.
21. Subject has life expectancy < 2 years.
22. Subject is, in the opinion of the Investigator or designee, unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason. This includes completion of Subject Reported Outcome instruments.
23. Subject is currently participating in another clinical investigation (except for non-invasive observational studies) that has not yet completed its primary endpoint.
24. Subject intends to participate in another investigational drug or device clinical investigation (except for non-invasive observational studies) within 12 months after the index procedure.
25. Subject has other medical illness (e.g., cancer or congestive heart failure) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy less than 2 years.
26. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
27. Subject has active symptoms and/or a positive test result of COVID-19 or other rapidly spreading novel infectious agent within the prior 2 months.

Angiographic Exclusion Criteria:

1. Target lesion/vessel meets any of the following criteria:

   * Prevents complete angioplasty balloon (plain old balloon angioplasty [POBA], scoring balloon, or cutting balloon) inflation, such as:

     * Heavy calcified lesion
     * Requires additional device for lesion preparation (e.g. rotablator or laser).
   * Anatomy proximal to or within the lesion that prevents proper placement of delivery system:

     * Extreme angulation (≥ 90°) proximal to or within the target lesion.
     * Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion.
   * Involves a bifurcation of which the side branch will be jailed by the struts and requiring side branch pre-dilatation by Kissing Balloon Technique, and/or stenting
   * Is located:

     * In left main or there is a ≥30% diameter stenosis in the left main (unless the left main lesion is a protected left main (i.e. a patent bypass graft to the left anterior descending coronary artery [LAD] and/or left circumflex coronary artery [LCX] arteries is present), and there is no intention to treat the protected left main lesion.
     * Within 3 mm of the origin of the LAD or LCX.
     * Within 3 mm of aorto-ostial right coronary artery (RCA).
     * In a bypass graft or distal to anastomotic site of bypass graft.
   * With total occlusion (TIMI flow 0), prior to crossing with the wire.
   * Contains thrombus
   * The subject has been previously treated with a stent within 1-year prior to the index procedure such that the ABT NG DES 48 would need to cross the stent to reach the target lesion.
2. Unsuccessful target lesion pre-dilatation, defined as the presence of one or more of the following:

   * Failed for a full inflation of the pre-dilatation balloon.
   * TIMI flow grade <3 (per visual estimation).
   * Any angiographic complication (e.g. distal embolization, no-reflow)
   * Any dissection National Heart, Lung, and Blood Institute (NHLBI) grade D-F.
   * Any chest pain lasting > 5 minutes.
   * Any ST-segment depression or elevation lasting > 5 minutes.
   * Side branch requires additional dilatation/stenting caused by plaque shift, carina shift or may require additional dilatation/stenting after stent implantation, per the operator's assessment.
3. Non-target lesion meets any of the following criteria:

   * Is located in the target vessel
   * Is located in the left main location
   * Is restenotic from a previous stent implantation
   * Is located within a saphenous vein graft or an arterial graft
   * Is with a TIMI flow 0 (total occlusion) prior to guide wire crossing
   * Involves a complex bifurcation that needs two-stent strategy.
4. Treatment of non-target lesion is not deemed successful.

Note: A successful treatment is defined as a treatment resulted in a mean lesion diameter stenosis < 30% in 2 near-orthogonal projections with TIMI 3 flow, as visually assessed by the physician, without the occurrence of prolonged chest pain or ECG changes consistent with MI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2023-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Jen Chang, MD, Principal Investigator — Chang Gung Memorial Hospital; Ki E Park, MD, Principal Investigator — University of Florida/Malcom Randall VAMC
Locations (25):
- United States (18):
  - HonorHealth, Scottsdale, Arizona
  - Scripps Memorial Hospital - La Jolla, La Jolla, California
  - UCLA Medical Center Santa Monica, Santa Monica, California
  - The Cardiac & Vascular Institute Research Foundation, LLC, Gainesville, Florida
  - Shands at the University of Florida, Gainesville, Florida
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Patrick Hospital, Missoula, Montana
  - Mount Sinai Hospital, New York, New York
  - The Lindner Center, Cincinnati, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Pinnacle Health System, Harrisburg, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Baylor Scott & White Heart & Vascular Hospital, Dallas, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
- Australia (3):
  - Liverpool Hospital, Liverpool, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal North Shore Hospital, St Leonards
- Taiwan (4):
  - Chang Gung Memorial Hospital, Linkou District, North Taiwan
  - National Taiwan University Hospital, Taipei, North Taiwan
  - Cheng Hsin General Hospital, Taipei, North Taiwan
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, South Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 107 subjects were registered at 25 study sites globally. Of the 107 registered subjects, the study device was successfully implanted in 105 subjects and 2 subjects were excluded from analyses as they did not receive the study device implanted. The study registered the first subject on June 17, 2020, and the last subject on September 17, 2021. The last 1-year follow-up visit occurred on October 7, 2022. The last 2-year follow-up visit occurred on September 18, 2023.
Pre-assignment Details: One subject expired during the 2-year-follow up window and is showing as "completed" under overall study status.
Period: Overall Study
Arm/Group | ABT NG DES 48 EECSS
Started | 105
Completed | 96
Not Completed | 9
Not completed — Death | 7
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABT NG DES 48 EECSS
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 102
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 62
  More than one race | 0
  Unknown or Not Reported | 4
Hypertension [Count of Participants; unit: Participants] | 87
Dyslipidemia [Count of Participants; unit: Participants] | 93

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of 1-Year Target Lesion Failure (TLF)
Description: Target Lesion Failure (TLF) is defined as the composite rate of cardiac death (CD), target vessel myocardial infarction [TV-MI] (per SCAI MI definition), and clinically indicated target lesion revascularization [CI-TLR])
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: Percentage of events
Arm/Group | ABT NG DES 48 EECSS
Number analyzed (Participants) | 105
Percentage of events | 5.7
Statistical Analysis 1: Comparison: ABT NG DES 48 EECSS; Test type: Superiority; p < 0.0001, Z test using Kaplan Meier survival estim

2. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: In-hospital 6 to 12 hours post procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | ABT NG DES 48 EECSS
Number analyzed (Participants) | 105
participants
  Target Lesion Failure per SCAI definition | 4
  Target Lesion Failure per ARC 2 definition | 5
  Target Lesion Failure per 4th Universal definition | 3

3. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | ABT NG DES 48 EECSS
Number analyzed (Participants) | 105
participants
  Target Lesion Failure per SCAI definition | 5
  Target Lesion Failure per ARC 2 definition | 6
  Target Lesion Failure per 4th Universal definition | 4

4. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 180 days
Population: Subjects who were truly lost-to-follow-up, defined as subjects who are terminated through a given time point without any DMR events (all death, all MI regardless of MI definition, all revascularization), were removed from the TLF analysis at specific time point. One subject withdrew from the study prior to 6 month (180 days) post procedure. Subject number analyzed at 180 days time frame went down from 105 to 104.
Measure: Number; unit: participants
Arm/Group | ABT NG DES 48 EECSS
Number analyzed (Participants) | 104
participants
  Target Lesion Failure per SCAI definition | 5
  Target Lesion Failure per ARC 2 definition | 6
  Target Lesion Failure per 4th Universal definition | 4

5. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 1 year
Population: Subjects who are terminated through a given time point without any DMR events were removed from TLF analysis at specific time point.
  One subject withdrew from the study prior to 6 month (180 days) post procedure, the subject number analyzed went down from 105 to 104.
  At 391 days after enrollment (within 1 year follow up window), one subject withdrew from the study, the subject was included in TLF analysis at 1 year, subject number analyzed at 1 year time frame stayed at 104.
Measure: Number; unit: participants
Arm/Group | ABT NG DES 48 EECSS
Number analyzed (Participants) | 104
participants
  Target Lesion Failure per SCAI definition | 6
  Target Lesion Failure per ARC 2 definition | 7
  Target Lesion Failure per 4th Universal definition | 5

6. Secondary Outcome: Number of Participants With Target Lesion Failure (TLF)
Description: as for outcome 1
Time Frame: 2 year
Population: Subjects who are terminated through a given time point without any DMR events were removed from TLF analysis at specific time point.
  1 subject withdrew from the study prior to 6 month (180 days) post procedure, subject number went down from 105 to 104.
  At 391 days after enrollment (within 1 year follow up window), one subject withdrew from the study was included in TLF analysis at 1 year and excluded from 2 year time frame, hence number analyzed at 2 year time frame went down from 104 to 103.
Measure: Count of Participants; unit: Participants
Arm/Group | ABT NG DES 48 EECSS
Number analyzed (Participants) | 103
Participants
  Target Lesion Failure per SCAI definition | 9
  Target Lesion Failure per ARC 2 definition | 10
  Target Lesion Failure per 4th Universal definition | 8

ADVERSE EVENTS:
Time Frame: 2 Year
Arm/Group | ABT NG DES 48 EECSS
All-Cause Mortality (participants affected / at risk) | 8/105
Serious Adverse Events (participants affected / at risk) | 42/105
Other Adverse Events (participants affected / at risk) | 49/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT NG DES 48 EECSS (N=105)
ANAEMIA (Blood and lymphatic system disorders) | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 8
ARRHYTHMIA (Cardiac disorders) | 5
ATRIAL FIBRILLATION (Cardiac disorders) | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 7
CORONARY ARTERY DISSECTION (Cardiac disorders) | 2
MYOCARDIAL INFARCTION (Cardiac disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
CHEST PAIN (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 1
CORONA VIRUS INFECTION (Infections and infestations) | 1
URINARY TRACT INFECTION (Infections and infestations) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
PLAQUE SHIFT (Injury, poisoning and procedural complications) | 1
COLONOSCOPY (Investigations) | 1
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 2
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 3
DYSTONIA (Nervous system disorders) | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 3
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1
HAEMORRHAGE (Vascular disorders) | 4
HYPOTENSION (Vascular disorders) | 3
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1
ANGINA UNSTABLE (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
ASTHENIA (General disorders) | 1
DEATH (General disorders) | 4
NON-CARDIAC CHEST PAIN (General disorders) | 1
ORAL CANDIDIASIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 2
SEPSIS (Infections and infestations) | 2
BLOOD CULTURE POSITIVE (Investigations) | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
COMA (Nervous system disorders) | 1
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2
FINGER AMPUTATION (Surgical and medical procedures) | 1
AORTIC ANEURYSM (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABT NG DES 48 EECSS (N=105)
NON-CARDIAC CHEST PAIN (General disorders) | 9
CARDIAC ENZYMES INCREASED (Investigations) | 38
CORONA VIRUS INFECTION (Infections and infestations) | 8
DIZZINESS (Nervous system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/48/NCT04282148/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT04282148/SAP_001.pdf